CLINICAL TRIAL: NCT04892667
Title: Early Detection of Patients at Risk of Developing Anthracycline Cardiotoxicity With TEP/CT -FDG
Acronym: DETECT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: APHP191102; IDRCB 2020-A01971-38 (Other: ANSM)
Record Dates: First submitted 2021-04-13; First posted 2021-05-19 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Lymphoma, Non-Hodgkin; Lymphoma, Hodgkin
Keywords: Lymphoma; Anthracyclines; Cardiac toxicity; Chemotherapy; Left Ventricular Systolic Dysfunction (LVSD); 18F-FDG; Echocardiography; PET-CT; Strain longitudinal global (SLG)
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Hodgkin Disease; Lymphoma; Cardiotoxicity; Ventricular Dysfunction, Left | interventions — Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients with lymphoma (Hodgkin's or non Hodgkin's) (Other)
  Interventions: Other: Intervention

INTERVENTIONS:
Other: Intervention — Evaluation of the sensitivity of the cardiac uptake of 18F-FDG measured on D28 +/- 7 days, D42 +/- 7 days ou D56 + 4 days of the administration of ATCs to identify at 1 year the patients at risk of occurrence of a LVSD defined by a drop of more than 10 units of the LVEF and LVEF < 53%.
  The patient participating in the study needs to respect a minimum of 12-hour fasting period, a high protein and a low-carbohydrate diet prior to performing PET/CT in order to limit physiological 18F-FDG myocardial fixation.

SUMMARY:
Management of patients with lymphoma is based on the administration of a chemotherapy containing anthracyclines (ATC), and allows cure rates of 65% to 80% at 5 years. The administration of ATCs can lead to an increase in the risk of the Left Ventricular Systolic dysfunction (LVSD) which ranges from 6 to 15% at 1 year, and of heart failure from which impact at 3.5 years can reach 5%. The major issue in the management of this toxicity is the early identification of this population for monitoring and prevention. No pharmacological intervention strategy is currently recommended.

According to the recommendations of the European Society of Cardiology, this identification is based on the measurement of the left ventricular ejection fraction (LVEF) and the overall longitudinal strain (SLG) before and after the last administration of ATC ( at D84 or D126, depending on the duration of the chemotherapy protocol). Recent studies have evaluated the diagnostic performance of earlier strategies highlighting the benefit of SLG measured after 150 mg / m2 of ATC (D28 +/- 7 days, D42 +/- 7 days ou D56 + 4 days). However, the tools are lacking to detect these patients as close as possible to the onset of ATC, a necessary condition for effective secondary prevention. The hypothesis is that an early assessment of myocardial binding of 18F-FDG, analyzed during the first routine PET / CT scan as part of the assessment of the response to chemotherapy (D28 +/- 7 days, D42 +/- 7 days ou D56 + 4 days) should verify a population at risk of developing LVSD at 1 year.

DETAILED DESCRIPTION:
This is a study that evaluates the sensitivity of the cardiac uptake of 18F-FDG measured on D28 +/- 7 days, D42 +/- 7 days ou D56 + 4 days of the administration of ATCs to identify at 1 year the patients at risk of occurrence of a LVSD defined by a drop of more than 10 units of the LVEF and LVEF <53%.

Design : A multicenter clinical trial with 11 sites participating in the study.

Sample size : 484 patients

Duration of inclusion: 37 months Patient observation period: 12 months Total duration: 49 months

Assessment :

There is an inclusion visit, then protocol visits at D28 +/- 7 days, D42 +/- 7 days ou D56 + 4 days, D84 or D126 and at the end of the study (M12).

There is no interim analysis planned. Analyzes will be performed at the end of the test after reviewing the data and freezing the database.

ELIGIBILITY:
Inclusion Criteria:

* Patients of at least 18 years of age, treated as part of an initial extension assessment (staging) of a lymphoma (Hodgkin's or non-Hodgkin's)
* Treatment with a chemotherapy protocol containing Anthracyclines (ABVD protocol, enhanced BEACOPP, R CHOP, CHOP, CHOEP, EPOCH, ACVBP)
* Signed informed consent
* Affiliation to a social security system (AME excepted)

Exclusion Criteria:

* FEVG<53%
* Cardiological symptomatic patient (Dyspnea, angina, palpitations, syncope, left ventricular insufficiency, right ventricular insufficiency, overall heart failure)
* Patient for whom PET/CT invalidates the presence of lymphoma (Hodgkin's or non-Hodgkin's)Uncontrolled blood pressure (AP) (systolic AP > 140 mm Hg and/or diastolic AP > 90 mmHg)
* Myocardial infarction in the 3 months prior to inclusion
* Heart failure in the 3 months prior to inclusion
* Severe symptomatic or asymptomatic mitral valvulopathy
* Symptomatic or asymptomatic tight aortic stenosis
* Atrial Fibrillation
* Pregnant or lactating woman
* Hypersensitivity to 18F-FDG
* Patient under guardianship or curatorship
* Patient under State Medical Aid

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2026-03-17 (Estimated); Study Completion 2026-03-17 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the cardiac uptake of 18F-FDG | Day 28 +/- 7 days, Day 42 +/- 7 days or Day 56 + 4 days
  Evaluation of the cardiac uptake of 18F-FDG measured on Day 42 of the administration of ATCs to identify at 1 year the patients at risk of occurrence of a LVSD defined by a drop of more than 10 units of the LVEF and LVEF <53%.

SECONDARY OUTCOMES:
The specificity, the negative predictive value and the positive predictive value of 18F-FDG cardiac uptake | Day 28 +/- 7 days, Day 42 +/- 7 days or Day 56 + 4 days
  Evaluate the specificity, the negative predictive value and the positive predictive value of 18F-FDG cardiac uptake of ATC administration to identify patients at risk of developing LVSD at 1 year (defined by a decrease of more than 10 units of LVEF and LVEF &amp;amp;amp;amp;amp;lt; 53%).
Evaluate with the echocardiography performed at the end of chemotherapy the sensitivity, specificity, the negative predictive value and the positive predictive value of the SLG change (difference of | Day 84 and Day 126
  SLG change is defined as: difference in SLG measured prior to chemotherapy administration and at the end of chemotherapy (Day 84 or Day 126 depending on the chemotherapy protocol) .
Compare PET/CT sensitivities at D28 +/- 7 days, D42 +/- 7 days or D56 + 4 days and SLG variation between the start and the end of chemotherapy administration (D84 or D126 depending on the chemotherapy protocol) to identify patients at risk of LVSD at 1 y | Day 28 +/- 7 days, Day 42 +/- 7 days or Day 56 + 4 days
Search for an intensity threshold in Standard Uptake Value (SUV)) of global 18F-FDG uptake to predict the occurrence of LVSD at 1 year. | 1 year
Evaluate the concordance between the result of the 18F-FDG cardiac uptake performed at D28 +/- 7 days, D42 +/- 7 days or D56 + 4 days assessed by the investigator and the result obtained at the centralized review. | Day 28 +/- 7 days, Day 42 +/- 7 days or Day 56 + 4 days

CONTACTS AND LOCATIONS:
Overall Officials: Stephane EDERHY, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Cardiology department, Paris, France